CLINICAL TRIAL: NCT00048048
Title: An Open-label, Randomized, Multi-centre, Multiple Dose Trial to Investigate the Efficacy and Safety of Subcutaneous Injections of RO0503821 at Different Dosing Intervals in Patients With Chronic Renal Anemia Who Are Not on Renal Replacement Therapy
Brief Title: A Study of Mircera in Anemic Patients With Chronic Kidney Disease Not Yet on Dialysis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16528
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (9):
- Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) (Experimental): Eligible participants will be receiving RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) at a dose of 0.15 microgram per kilogram (mcg/kg) subcutaneously (SC) once every week to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 2 (RO0503821, 0.3 mcg/kg 1x/Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 0.3 mcg/kg SC once every week to complete the dosage of 1.8 mcg/kg up to 6 weeks (Week 7 to Week 12). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 0.6 mcg/kg SC once every week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 0.3 mcg/kg SC once every two week, to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 0.6 mcg/kg SC once every two week, to complete the dosage of 1.8 mcg/kg up to 6 weeks (Week 7 to Week 12). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 1.2 mcg/kg SC once every two week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 0.45 mcg/kg SC once every three week, to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 0.9 mcg/kg SC once every three week, to complete the dosage of 1.8 mcg/kg up to 6 weeks (Week 7 to Week 12). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Cohort 9 (RO0503821,1.8 mcg/kg 1x/3 Week) (Experimental): Eligible participants will be receiving RO0503821 at a dose of 1.8 mcg/kg SC once every three week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants will be followed-up for one week post the treatment period. During extension Years 1 and 2, the participants will remain at the same frequency of administration as that of core treatment period.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — Differing doses and frequencies of sc administration

SUMMARY:
This study will evaluate the efficacy and safety of different subcutaneous starting doses and dosing frequencies of Mircera in anemic patients with chronic kidney disease not yet on dialysis. The anticipated time on study treatment is 3-12 months and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* not receiving renal replacement therapy.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* administration of any investigational drug within 30 days preceding the screening visit and during the run-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2002-03; Primary Completion 2003-10 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (5):
  - Birmingham, Alabama
  - San Diego, California
  - Detroit, Michigan
  - Las Vegas, Nevada
  - Portland, Oregon
- Canada (2):
  - Edmonton, Alberta
  - Vancouver, British Columbia
- Mexico (2):
  - Mexico City
  - Monterrey
- Poland (3):
  - Gdansk
  - Krakow
  - Wroclaw
- United Kingdom (2):
  - Belfast
  - London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 15 centers in 5 countries from 07 March 2002 until 23 November 2004 (last date of extension Year 2)
Groups:
- Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week): Eligible participants received RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) at a dose of 0.15 microgram per kilogram (mcg/kg) subcutaneously (SC) once every week to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 2 (RO0503821, 0.3 mcg/kg 1x/Week): Eligible participants received RO0503821 at a dose of 0.3 mcg/kg SC once every week to complete the dosage of 1.8 mcg/kg up to 6 weeks (Week 7 to Week 12). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week): Eligible participants received RO0503821 at a dose of 0.6 mcg/kg SC once every week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week): Eligible participants received RO0503821 at a dose of 0.3 mcg/kg SC once every two week, to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week): Eligible participants received RO0503821 at a dose of 0.6 mcg/kg SC once every two week, to complete the dosage of 1.8 mcg/kg up to 6 weeks (Week 7 to Week 12). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week): Eligible participants received RO0503821 at a dose of 1.2 mcg/kg SC once every two week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week): Eligible participants received RO0503821 at a dose of 0.45 mcg/kg SC once every three week, to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week): Eligible participants received RO0503821 at a dose of 0.9 mcg/kg SC once every three week, to complete the dosage of 1.8 mcg/kg up to 6 weeks (Week 7 to Week 12). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 9 (RO0503821, 1.8 mcg/kg 1x/3 Week): Eligible participants received RO0503821 at a dose of 1.8 mcg/kg SC once every three week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- RO0503821 (1x/Week): Eligible participants received RO0503821 at the dose of either 0.15 mcg/kg (Cohort 1) or 0.3 mcg/kg (Cohort 2) or 0.6 mcg/kg (Cohort 3) SC once weekly over a period of 18 weeks. Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- RO0503821 (1x/2Week): Eligible participants received RO0503821 at the dose of either 0.3 mcg/kg (Cohort 4) or 0.6 mcg/kg (Cohort 5) or 1.2 mcg/kg (Cohort 6) SC once every two weeks over a period of 18 weeks. Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- RO0503821 (1x/3week): Eligible participants received RO0503821 at the dose of either 0.45 mcg/kg (Cohort 7) or 0.9 mcg/kg (Cohort 8) or 1.8 mcg/kg (Cohort 9) SC once every three weeks over a period of 18 weeks. Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
Period: Core Treatment
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821, 0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821, 1.8 mcg/kg 1x/3 Week) | RO0503821 (1x/Week) | RO0503821 (1x/2Week) | RO0503821 (1x/3week)
Started | 6 | 6 | 10 | 6 | 6 | 9 | 6 | 6 | 10 | 0 | 0 | 0
Completed | 6 | 6 | 9 | 6 | 6 | 9 | 6 | 5 | 10 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Extension Year 1
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821, 0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821, 1.8 mcg/kg 1x/3 Week) | RO0503821 (1x/Week) | RO0503821 (1x/2Week) | RO0503821 (1x/3week)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 (Participants (Cohorts 1, 2, and 3) who completed core, entered extension period (entry optional).) | 16 (Participants (Cohorts 4, 5, and 6) who completed core, entered extension period (entry optional).) | 19 (Participants (Cohorts 7, 8, and 9) who completed core, entered extension period (entry optional).)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Not completed — Early withdrawals | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Period: Extension Year 2
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821, 0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821, 1.8 mcg/kg 1x/3 Week) | RO0503821 (1x/Week) | RO0503821 (1x/2Week) | RO0503821 (1x/3week)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Twelve participants who completed Extension Year 1 were switched to RO0503821 (1x/2Week).) | 23 (A portion of participants who completed Extension Year 1 + 12 participants from RO0503821 (1X/Week).) | 15 (A portion of participants who completed Extension Year 1, entered Extension Year 2 (entry optional).)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 19 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Early withdrawals | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Population: The safety population was considered for analysis which included all participants who received at least one dose of study drug.
Groups:
- Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week): Eligible participants received RO0503821 at a dose of 0.15 mcg/kg SC once every week to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 2 (RO0503821,0.3 mcg/kg 1x/Week): Eligible participants received RO0503821 at a dose of 0.3 mcg/kg SC once every week to complete the dosage of 1.8 mcg/kg up to 6 weeks (Week 7 to Week 12). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 3 (RO0503821,0.6 mcg/kg 1x/Week): Eligible participants received RO0503821 at a dose of 0.6 mcg/kg SC once every week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 9 (RO0503821,1.8 mcg/kg 1x/3 Week): Eligible participants received RO0503821 at a dose of 1.8 mcg/kg SC once every three week, to complete the dosage of 3.6 mcg/kg up to 6 weeks (Week 13 to Week 18). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821,0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821,0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821,1.8 mcg/kg 1x/3 Week) | Total
Number analyzed (Participants) | 6 | 6 | 10 | 6 | 6 | 9 | 6 | 6 | 10 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (21.66) | 70.0 (13.75) | 58.0 (16.55) | 60.3 (16.80) | 62.7 (21.29) | 62.3 (12.63) | 66.5 (9.42) | 54.5 (16.85) | 58.3 (18.42) | 60.9 (16.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 6 | 4 | 5 | 6 | 4 | 5 | 4 | 42
  Male | 2 | 2 | 4 | 2 | 1 | 3 | 2 | 1 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Change in Hemoglobin Over Time Between Baseline and End of Initial Treatment Based on Individual Regression Slopes
Description: The primary efficacy variable was blood Hb level and its changes from Baseline (defined as the mean Hb of Screening assessment (SA) (Week -3), Weeks -2 and -1 of the Run-in period) over time during the core treatment period. For each participant, the primary efficacy parameter was the change in hemoglobin level over time based on regression slopes. All values until end-of-initial treatment (EOIT), defined as the last observed value before a dose change or blood transfusion, were included in the calculation of this endpoint. For participants without any dose adjustments, the EOIT value was identical to the value for Week 19.
Time Frame: From Baseline (Day -28 to Day 1) to EOIT (Week 19)
Population: The Intent-to-Treat (ITT) population was defined as all randomized participants. Maximum number of participants with available data was reported.
Measure: Median (Inter-Quartile Range); unit: gram/deciliter (g/dL)
Groups:
- Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week): Eligible participants in received RO0503821 at a dose of 0.15 mcg/kg SC once every week to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week): Eligible participants in received RO0503821 at a dose of 0.3 mcg/kg SC once every two week, to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
- Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week): Eligible participants in received RO0503821 at a dose of 0.45 mcg/kg SC once every three week, to complete the dosage of 0.9 mcg/kg up to 6 weeks (Week 1 to Week 6). Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821, 0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821, 1.8 mcg/kg 1x/3 Week)
Number analyzed (Participants) | 6 | 6 | 10 | 6 | 6 | 9 | 6 | 6 | 10
gram/deciliter (g/dL) | 0.48 [-0.23 to 1.23] | 1.08 [0.98 to 1.32] | 1.34 [0.47 to 2.12] | 0.17 [-0.47 to 0.52] | 0.27 [-0.47 to 1.11] | 2.17 [1.38 to 2.61] | 0.41 [0.27 to 0.73] | 0.83 [0.03 to 1.75] | 1.28 [0.86 to 1.67]
Statistical Analysis 1: Comparison: Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) vs Cohort 2 (RO0503821, 0.3 mcg/kg 1x/Week) vs Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week); All cohorts with dosing frequency 1X/ Week; Test type: Superiority or Other; Least square mean = 0.979, 95% CI 2-sided [0.534 to 1.425], Standard Error of Mean 0.223 — To analyze the appropriateness of the chosen conversion factors, a second regression analysis was carried out. This regression was on the three conversion factor dose groups, using the regression slope estimates of Hb. This was not pre-specified
Statistical Analysis 2: Comparison: Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) vs Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) vs Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week); All cohorts with dosing frequency 1X/ 2Week; Test type: Superiority or Other; Least square mean = 0.851, 95% CI 2-sided [0.395 to 1.307], Standard Error of Mean 0.228 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) vs Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) vs Cohort 9 (RO0503821, 1.8 mcg/kg 1x/3 Week); All cohorts with dosing frequency 1X /3 Week; Test type: Superiority or Other; Least square mean = 0.932, 95% CI 2-sided [0.488 to 1.377], Standard Error of Mean 0.222 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Hematocrit Levels at End of Initial Treatment Under Constant Dosing Regimen
Description: Hematocrit (Hct) levels at end of initial treatment under constant dosing regimen were reported. Baseline (Day -28 to Day 1) Hct values was calculated as the mean of the SA (Week -3) and Run-in period (Weeks -2 and -1). For all participants, an EOIT value was calculated as the last observed Hct value before a dose change or blood transfusion. For participants without any dose adjustments, the EOIT value was identical to the value for Week 19.
Time Frame: From Baseline (Day -28 to Day 1) to EOIT (Week 19)
Population: The ITT population was defined as all randomized participants. Maximum number of participants with available data was reported.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821,0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821,0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821,1.8 mcg/kg 1x/3 Week)
Number analyzed (Participants) | 6 | 6 | 10 | 6 | 6 | 9 | 6 | 6 | 10
g/dL | 31.10 [30 to 33.10] | 39.10 [32.70 to 39.90] | 36.95 [32.30 to 42] | 28.40 [28 to 31.90] | 34.70 [32 to 37.70] | 40.50 [34.40 to 42.20] | 32.70 [27.70 to 32.90] | 37.75 [26.60 to 39.00] | 39 [33.90 to 42.30]

3. Secondary Outcome: Reticulocyte Count at End of Initial Treatment Under Constant Dosing Regimen
Description: Reticulocyte levels at EOIT under constant dosing regimen was analysed and reported. Baseline (Day -28 to Day 1) reticulocyte values were calculated as the mean of the SA (Week -3) and Run-in period (Weeks -2 and -1). For all participants, an EOIT value was calculated as the last observed reticulocyte count before a dose change or blood transfusion. For participants without any dose adjustments, the EOIT value was identical to the value for Week 19.
Time Frame: From Baseline (Day -28 to Day 1) to EOIT (Week 19)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Cells x10^3/UL
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821,0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821,0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821,1.8 mcg/kg 1x/3 Week)
Number analyzed (Participants) | 3 | 6 | 10 | 5 | 6 | 9 | 5 | 6 | 10
Cells x10^3/UL | 71.80 [45.0 to 89.70] | 46.30 [42.00 to 50.00] | 44.70 [36.56 to 72.50] | 51.80 [48.30 to 54.20] | 72.80 [39.0 to 90.0] | 59.20 [40.90 to 63.50] | 25.20 [20.0 to 43.0] | 38.45 [28.60 to 50.90] | 56.20 [39.70 to 70.00]

4. Secondary Outcome: Number of Participants With Any Serious Adverse Events and Any Adverse Events
Description: An Adverse Events (AEs) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious Adverse Events (SAEs) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes. The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time all results for the two long term safety periods were displayed by dose schedule group only.
Time Frame: Up to Week 125
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/Week) | RO0503821 (1x/2Week) | RO0503821 (1x/3week)
Number analyzed (Participants) | 22 | 21 | 22
participants
  Participants with SAEs | 11 | 9 | 12
  Participants with AEs | 22 | 21 | 22

5. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities for Blood Chemistry and Electrolytes Over Time
Description: Marked abnormality was defined as above and/or below a value (according to the Roche specified limits) which was considered to be potentially clinically relevant. The Roche reference range are: white blood cells (WBC) (3.0-18.0 10^9 cells/L), platelets (100-550 10^9 cells/L), alanine aminotransferase (ALT) [0-110 units per litre (U/L)], alkaline phosphatase (ALP) (0-220 U/L), aspartate aminotransferase (AST) (0-80 U/L), albumin >= 30 g/L, phosphate [0.75 - 1.60 millimoles per liter (mmol/L)], potassium (2.9 - 5.8 mmol/L), total bilirubin (0-17 µmol/L), lymphocytes (1- 4.80 10^9 cells/L), eosinophils (0 - 0.45 10^9 cells/L), monocytes (0 - 0.8 10^9 cells/L), and neutrophils (1.80 - 7.70 10^9 cells/L). The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time, all results for the two long term safety periods were displayed by dose schedule group only.
Time Frame: Up to Week 125
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/Week) | RO0503821 (1x/2week) | RO0503821 (1x/3week)
Number analyzed (Participants) | 22 | 21 | 22
participants
  Platelets - High, n = 16, 15, 19 | 0 | 1 | 0
  Platelets - Low, n = 16, 15, 19 | 0 | 0 | 3
  WBC - High, n = 16, 15, 19 | 0 | 0 | 1
  Eosinophils - High, n = 15, 15, 19 | 0 | 1 | 2
  Lymphocytes - Low, n = 15, 15, 19 | 2 | 2 | 1
  Monocytes - High, n = 15, 15, 19 | 0 | 0 | 1
  Neutrophils - High, n = 15, 15, 19 | 0 | 3 | 3
  Neutrophils - Low, n = 15, 15, 19 | 0 | 2 | 0
  ALT - High, n = 22, 21, 22 | 1 | 1 | 1
  ALP - High, n = 22, 21, 22 | 1 | 0 | 2
  AST - High, n = 22, 21, 22 | 2 | 1 | 2
  Total bilirubin - High, n = 22, 21, 22 | 0 | 0 | 1
  Albumin - Low, n = 22, 21, 22 | 2 | 0 | 2
  Phosphate - High , n = 12, 13, 14 | 7 | 6 | 1
  Phosphate - Low, n = 12, 13, 14 | 2 | 1 | 1
  Potassium - High, n = 22, 21, 22 | 3 | 2 | 2
  Potassium - Low, n = 22, 21, 22 | 1 | 0 | 0

6. Secondary Outcome: Heart Rate Over Time
Description: Heart rate was defined as the measure of heart beats per minute (bpm). The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time all results for the two long term safety periods were displayed by dose schedule group only.
Time Frame: Up to Week 125
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- RO0503821 (1x/3week): Eligible participants received RO0503821 at the dose of either 0.45 (Cohort 7) or 0.9 mcg/kg (Cohort 8) or 1.8 mcg/kg (Cohort 9) SC once every three weeks over a period of 18 weeks. Participants were followed-up for one week post the treatment period. During extension Years 1 and 2, the participants remained at the same frequency of administration as that of core treatment period.
Arm/Group | RO0503821 (1x/Week) | RO0503821 (1x/2week) | RO0503821 (1x/3week)
Number analyzed (Participants) | 22 | 21 | 22
bpm | 65.6 (4.3) | 68.4 (9.8) | 75.4 (10.4)

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure
Description: Change from Baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) is calculated as the end of treatment values minus the Baseline value. Baseline (Day -28 to Day 1) values were calculated as the mean of the SA (Week -3) and Run-in period (Week -2 and Week -1).
Time Frame: From Baseline (Day -28 to Day 1) to Week 125
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1 (RO0503821, 0.15 mcg/kg 1x/Week) | Cohort 2 (RO0503821,0.3 mcg/kg 1x/Week) | Cohort 3 (RO0503821, 0.6 mcg/kg 1x/Week) | Cohort 4 (RO0503821, 0.3 mcg/kg 1x/2 Week) | Cohort 5 (RO0503821, 0.6 mcg/kg 1x/2Week) | Cohort 6 (RO0503821, 1.2 mcg/kg 1x/2 Week) | Cohort 7 (RO0503821, 0.45 mcg/kg 1x/3 Week) | Cohort 8 (RO0503821, 0.9 mcg/kg 1x/3Week) | Cohort 9 (RO0503821,1.8 mcg/kg 1x/3 Week)
Number analyzed (Participants) | 6 | 6 | 10 | 6 | 6 | 9 | 6 | 6 | 10
mmHg
  DBP | 2 (10.5) | 5 (6.6) | 6 (5.9) | 6 (13.7) | 2 (9.4) | -3 (8.3) | 6 (10.3) | -2 (12.9) | 4 (10.3)
  SBP | 12 (20.2) | 2 (15.9) | 5 (16.7) | 2 (16.7) | 8 (3.8) | -11 (16.3) | 6 (16.5) | 3 (10.0) | -3 (25.5)

ADVERSE EVENTS:
Time Frame: Up to Week125
Description: SAEs and non SAEs are reported in safety analysis set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline. The study design tested 3 different starting dose conversion factors at 3 different dosing schedules during the core study period. As study drug doses can be modified continually over time all results for the two long term safety periods were displayed by dose schedule group only.
Arm/Group | RO0503821 (1x/Week) | RO0503821 (1x/2Week) | RO0503821 (1x/3week)
Serious Adverse Events (participants affected / at risk) | 11/22 | 9/21 | 12/22
Other Adverse Events (participants affected / at risk) | 16/22 | 18/21 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/Week) (N=22) | RO0503821 (1x/2Week) (N=21) | RO0503821 (1x/3week) (N=22)
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Prostatic disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Renal Cyst Ruptured (Renal and urinary disorders) | 2 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1
Bronchitis Acute (Infections and infestations) | 0 | 1 | 0
Clostridium Colitis (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 0 | 1
Vascular Pseudoaneurysm (Vascular disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/Week) (N=22) | RO0503821 (1x/2Week) (N=21) | RO0503821 (1x/3week) (N=22)
Urinary Tract Infection (Infections and infestations) | 3 | 4 | 5
Nasopharyngitis (Infections and infestations) | 1 | 4 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 2
Bronchitis Acute (Infections and infestations) | 0 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 2
Hepatitis C (Infections and infestations) | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 2
Oedema Peripheral (General disorders) | 1 | 5 | 3
Influenza Like Illness (General disorders) | 2 | 1 | 3
Fatigue (General disorders) | 0 | 3 | 0
Asthenia (General disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Renal Failure Chronic (Renal and urinary disorders) | 3 | 4 | 3
Renal Failure (Renal and urinary disorders) | 2 | 0 | 1
Hypertension (Vascular disorders) | 6 | 2 | 5
Gout (Metabolism and nutrition disorders) | 2 | 3 | 2
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperparathyroidism Secondary (Endocrine disorders) | 1 | 1 | 3
Hyperparathyroidism (Endocrine disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 3 | 3
Dizziness (Nervous system disorders) | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 6 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Angina Pectoris (Cardiac disorders) | 0 | 1 | 2
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Arteriovenous Fistula Operation (Surgical and medical procedures) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.